CLINICAL TRIAL: NCT06559189
Title: Phase I Dose Escalation and Preliminary Efficacy Study of Bispecific CD19 and CD22 Chimeric Antigen Receptor Co-Expressing T Cells (CD19x22 CAR T) in Pediatric Patients With Relapsed and/or Refractory B-Cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: CD19x22 Chimeric Antigen Receptor T-cell Therapy (CAR T) in Pediatric B-ALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0998.cc; NCI-2024-06242 (Other: CTRP)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Pediatric; Relapsed; Refractory; B-cell Acute Lymphoblastic Leukemia; Hematologic diseases
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Disease Burden Cohort (Experimental): ≥25% bone marrow lymphoblasts and/or non-CNS extramedullary disease. Dose escalation will proceed independently within each cohort using the Bayesian Optimal Interval (BOIN)design. Dose begins at DL -1(1x10^5 cells/kg).
  Interventions: Biological: CD19x22 CAR T
- Low Disease Burden Cohort (Experimental): <25% bone marrow lymphoblasts and no non-CNS extramedullary disease. Dose escalation will proceed independently within each cohort using the Bayesian Optimal Interval (BOIN)design. Dose begins at DL1 (3x10^5 cells/kg).
  Interventions: Biological: CD19x22 CAR T

INTERVENTIONS:
Biological: CD19x22 CAR T — The investigational product is an autologous, genetically modified CD19xCD22 CAR T cell product produced by the Gates Biomanufacturing Facility.

SUMMARY:
This study will evaluate the safety and tolerability of administering a novel bispecific CD19/CD22-directed CAR T cell product (CD19x22) for the treatment of relapsed or refractory pediatric B-ALL.

DETAILED DESCRIPTION:
This is an open-label Phase I trial consisting of 2 cohorts to determine the safety and tolerability of CD19x22 CAR T in Pediatric Patients with R/R B-ALL. This trial will include two parallel cohorts based on disease burden prior to lymphodepleting chemotherapy, Cohort 1: high disease burden cohort: defined as >=25% bone marrow lymphoblasts and/or non-CNS extramedullary disease, and Cohort 2: low disease burden cohort: defined as <25% bone marrow lymphoblasts and no non-CNS extramedullary disease. Dose escalation will proceed independently within each cohort using the Bayesian Optimal Interval (BOIN) design. This trial will enroll up to 53 patients with 21 patients in each cohort receiving treatment with lymphodepleting chemotherapy followed by CD19x22 CAR T cell infusion, with a total of up to 42 treated patients overall. Patients will be assessed for dose limiting toxicities (up to 28 days from infusion) to determine a maximum tolerated dose (MTD) and for preliminary efficacy through morphological remission rate and measurable residual disease (MRD) levels.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a history of B precursor ALL with any of the following conditions:

   1. Relapsed two or more times.
   2. Relapsed at any time after allogeneic bone marrow transplant (BMT).
   3. Relapse or refractory after single antigen targeting CAR T cell therapy.

   i. 90 days must have elapsed post previous CAR infusion prior to apheresis. d. Refractory to standard therapy as determined by the treating physician. e. Patient and/or parents declining BMT options and would prefer CAR T Therapy.
2. CD19 and/or CD22 present on last relapsed/refractory disease evaluation.
3. Performance score (Lansky or Karnofsky ≥ 50%; or Eastern Cooperative Oncology Group (ECOG) must be ≤2).
4. Meets criteria for potential leukapheresis collection or has leukapheresis product previously collected and stored per recommended guidelines.
5. Males OR non-pregnant, non-lactating females.
6. Aged 3 months to 30 years (inclusive) at time of consent and enrollment.
7. Provision of a signed and dated consent form from parent or guardian (patients < 18), the patient themselves (> 18), or legally authorized representative (patient > 18 who lack decision-making capacity) after standard of care (SOC) screening assessments are performed.
8. Stated willingness to comply with all study procedures and be available for the duration of the study.
9. Willingness to participate in long-term follow-up protocol.

Exclusion Criteria:

1. Active, uncontrolled central nervous system (CNS) leukemia that is progressive despite other therapies or leading to CNS symptoms (including but not limited to: seizures, paresis, aphasia, hemorrhage, dementia, psychosis, or movement disorders) as determined by the treating physician at eligibility, prior to lymphodepleting chemotherapy (LD chemo), and pre- CD19x22 CAR T cell infusion.
2. History of allogeneic stem cell transplantation prior to apheresis that meet the following criteria:

   1. Less than 100 days post-transplant;
   2. Evidence of active Graft-versus-Host Disease (GvHD) requiring systemic therapy;
   3. Less than 6 weeks post donor lymphocyte infusion (DLI).
3. Active, uncontrolled, life-threatening infection that at the determination of the treating physician would preclude safe apheresis or tolerance of lymphodepleting chemotherapy, cell infusion, or increased risk of cytokine release syndrome.
4. Evidence of severe organ dysfunction defined by:

   1. Baseline oxygen saturation of < 90% on room air
   2. Myocardial dysfunction (based on age standards): Ejection fraction ≤ 40% or shortening fraction ≤ 28%, evidence of physiologically significant pericardial effusion as determined by an echocardiogram (ECHO), and clinically significant electrocardiogram (ECG or EKG) findings
   3. Transaminases > 10x upper limit of normal (ULN) or bilirubin > 5x the ULN, unless thought to be related to primary disease
   4. Estimated Creatinine (Cr) clearance < 60 mL/min/1.73 m2 (if nuclear medicine GFR or other more specific testing exceeds this level than it can supersede the estimated clearance)
5. Subjects of childbearing or child-fathering potential that are not willing to practice birth control from the time of enrollment on this study and for 12 months after receiving the investigational product
6. Known HIV infection or active Hepatitis B or Hepatitis C infection.

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Safety Measured by Dose Limiting Toxicities (DLTs) | Infusion date to 28 days post-infusion
  The safety of the administering this bispecific CD19/CD22-directed CAR T cell product will be measured by assessing the DLTs in each disease burden cohort in a Bayesian optimal interval (BOIN) design to determine the MTD

SECONDARY OUTCOMES:
Overall Response Rate | 28 days post-infusion
  The efficacy of this bispecific CD19/CD22-directed CAR T cell product will be measured by evaluating the overall response rate in each disease burden stratum based on a morphologic disease assessment to measure bone marrow status at Day 28 post-infusion.
Minimal Residual Disease (MRD) Rate | Months 1, 2, 3, 6, 9, and 12
  The efficacy of this bispecific CD19/CD22-directed CAR T cell product will be monitored in each disease burden stratum by measuring peripheral blood MRD by next generation sequencing
Minimal Residual Disease (MRD) Rate | Months 1, 3, 6, and 12
  The efficacy of this bispecific CD19/CD22-directed CAR T cell product will be monitored in each disease burden stratum by measuring bone marrow MRD by flow cytometry and/or next generation sequencing.
CD19-Relapse | 1 year
  Cumulative incidence of CD19-relapse as determined by immunophenotype of leukemic blasts for subjects in each disease burden stratum will be calcualted using standard techniques using all enrolled patients and compared to published literature both from pre- and post-licensing clinical trials and/or reports.
Overall Survival | 1 year
  1-year overall survival (OS) rate in subjects with relapsed/refractory B-ALL treated with this bispecific CD19/CD22-directed CAR T cell product, stratified by disease burden.
Progression Free Survival | 1 year
  1-year progression-free survival (PFS) rate in subjects with relapsed/refractory B-ALL treated with this bispecific CD19/CD22-directed CAR T cell product, stratified by disease burden.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Fabrizio, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No